CLINICAL TRIAL: NCT04621539
Title: Validation of the Quick Sequential [Sepsis-related] Organ Failure Assessment (qSOFA) Predictive Model in the Prediction of Severe Infection - Sepsis in Obstetric Patients and Adverse Neonatal Outcomes: a Multicenter Study
Brief Title: Validation of the Quick Sequential [Sepsis-related] Organ Failure Assessment (qSOFA) in Obstetric Patients
Acronym: COLOSSAL
Status: Completed | Type: Observational
Sponsor: Fundación Grupo de Investigación en Cuidados Intensivos y Obstetricia (Other)
Responsible Party: Sponsor
Other Study IDs: 58259
Record Dates: First submitted 2020-10-08; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Severe Infection
Keywords: Sepsis; Pregnancy; qSOFA; Systemic Inflammatory Response Syndrome
MeSH Terms: conditions — Infections; Sepsis; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infected without an SMO: Defined as an acute infection not associated with admission to the intensive care unit (ICU), mechanical ventilation, or the use of vasopressors.
- Infected with an SMO: defined as an acute infection associated with intensive care unit (ICU) admission, mechanical ventilation, or vasopressor use.

SUMMARY:
Research problem: In 1991, the terms Systemic Inflammatory Response Syndrome (SIRS), severe sepsis, and septic shock were introduced, based on the pro-inflammatory theory, conforming to a list of classification criteria for each one. New criteria were recently created in search of coherence with the pathophysiological process that generates the infection in the host: SOFA and qSOFA scores. Neither of these two criteria has been standardized in the obstetric patient, taking into account the physiological alteration of many of the clinical and laboratory parameters that occur in pregnancy. The question that arises then is: Are the new sepsis criteria qSOFA and SOFA valid in comparison with the previous SIRS criteria for predicting adverse maternal and neonatal outcomes in obstetric patients diagnosed with infection? Aim: To evaluate the predictive model quick Sequential [Sepsis-related] Organ Failure Assessment (qSOFA) in comparison with the SIRS criteria for the prognosis of severe infection-sepsis in obstetric patients and adverse neonatal outcomes in different cities of Colombia.

Methodology: a longitudinal prospective cohort multicenter study will be carried out in selected centers in Colombia, with a data collection duration of at least 12 months. Data will be collected on clinical characteristics, health outcomes, and medical practices. Study participants will be followed during their stay at the health center. Follow-up will end at hospital discharge, transfer to a facility outside of participating geographic areas, or death. Neonates born to mothers included in the study will be followed until discharge from the hospital or 7 days after birth if they are still in the hospital, whichever comes first.

Expected results: This study seeks to evaluate the predictive model q SOFA and the prognosis of sepsis in obstetrics in comparison with the SIRS criteria, hoping to find that qSOFA is superior to the SIRS criteria for the identification of which obstetric patients diagnosed with an infection they will progress to sepsis and which patients with sepsis progress to septic shock, this would translate both at the maternal and neonatal level in a reduction of adverse events, prolonged stays, disabilities, sequelae, in addition to allowing preventive actions and control, which finally translate into protocols that allow better management of this entity.

ELIGIBILITY:
Inclusion Criteria:

* Patients in a state of pregnancy with a single fetus between 14 and 49 years old.
* Pregnant women (any gestational age) defined as a positive gravindex test and an obstetric ultrasound to prove it.
* Any suspected or confirmed infection during current hospital stay (primary admission or readmission) with or without organ dysfunction
* Any clinical signs suggestive of infection (eg, fever)
* Request for culture of body fluids (blood, urine, cerebrospinal fluid, etc.) or swab specimen (nasopharyngeal, oropharyngeal);
* Non-prophylactic use of antibiotics or other antimicrobials during admission or during hospital stay.
* Any health care related infection (eg, surgical site, episiotomy, IV, venipuncture, urinary catheterization, central line, etc.)
* Urinary tract infection of the lower urinary tract that requires hospitalization and in-hospital management for more than 48 hours.
* Herpes simplex, herpes zoster (shingles) with associated liver failure.

Note: observations on the inclusion criteria:

* Eligible women who remain in the health center for 12 hours or more, regardless of formal administrative admission, will be included in the study.
* Eligible women admitted or readmitted to a participating health center, regardless of length of hospital stay, will be included in the study.

Exclusion Criteria:

* Pregnant women of any age who do not sign the informed consent.
* Pregnant minors who do not sign the consent.
* Any non-serious or localized infection

  * Vaginosis, candidiasis
  * Fungal skin infections (athlete's foot, ringworm)
  * Otitis o Pharyngitis
* Any chronic uncomplicated infection

  * Sexually transmitted infections (gonorrhea, syphilis, Trichomonas, chlamydia, hepatitis, HIV).
  * Tuberculosis.
* Any colonization Microorganisms without clinical signs / symptoms)

  * Known vaginal, urethral and / or rectal colonization of group B beta-hemolytic streptococcus.
  * Asymptomatic bacteriuria
  * Known oropharyngeal colonization
* Patients with surgical wound infection other than caesarean section (hysterectomy, laparotomy or others)
* Any iatrogenic / hyperthermic hypothermia (eg related to epidural, thyroid storm, prostaglandin administration) during hospital stay.
* Use of any prescription of prophylactic antibiotics (eg, for colonization of beta-hemolytic streptococcus group B, after cesarean section, manual removal of the placenta, vaginal delivery);
* Patients referred from other institutions with more than 24 hours of management

Ages: 14 Years to 49 Years | Sex: Female
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Pregnant women, childbirth or within 42 days of termination of pregnancy, with infectious symptoms of any kind (obstetric - non-obstetric) who attend and are hospitalized in the selected clinics during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 2125 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
Admission to intensive care unit | 28 days
  need or admission to an intensive care unit
Use of vasopressors | 28 days
  use of vasoactive drugs (norepinephrine, epinephrine, vasopressin)
Prolonged ICU stay | 28 days
  Stay in intensive care unit for 72 hours

SECONDARY OUTCOMES:
Additional interventions | 28 days
  need for surgery (cesarean section - emergency hysterectomy, hysterectomy, chest tubes, etc.), invasive mechanical ventilation, use of arterial line, among others.

CONTACTS AND LOCATIONS:
Overall Officials: Carmelo R Dueñas-Castell, Msc, Principal Investigator — Gestion Salud IPS
Locations (1):
- Gestion Salud, Cartagena, Departamento de Bolívar, Colombia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Say L, Chou D, Gemmill A, Tuncalp O, Moller AB, Daniels J, Gulmezoglu AM, Temmerman M, Alkema L. Global causes of maternal death: a WHO systematic analysis. Lancet Glob Health. 2014 Jun;2(6):e323-33. doi: 10.1016/S2214-109X(14)70227-X. Epub 2014 May 5. PMID 25103301
- [Background] Surgers L, Valin N, Carbonne B, Bingen E, Lalande V, Pacanowski J, Meyohas MC, Girard PM, Meynard JL. Evolving microbiological epidemiology and high fetal mortality in 135 cases of bacteremia during pregnancy and postpartum. Eur J Clin Microbiol Infect Dis. 2013 Jan;32(1):107-13. doi: 10.1007/s10096-012-1724-5. Epub 2012 Aug 21. PMID 22907333
- [Background] Acosta CD, Bhattacharya S, Tuffnell D, Kurinczuk JJ, Knight M. Maternal sepsis: a Scottish population-based case-control study. BJOG. 2012 Mar;119(4):474-83. doi: 10.1111/j.1471-0528.2011.03239.x. Epub 2012 Jan 18. PMID 22251396
- [Background] Kankuri E, Kurki T, Carlson P, Hiilesmaa V. Incidence, treatment and outcome of peripartum sepsis. Acta Obstet Gynecol Scand. 2003 Aug;82(8):730-5. doi: 10.1034/j.1600-0412.2003.00265.x. PMID 12848644
- [Background] Bone RC, Balk RA, Cerra FB, Dellinger RP, Fein AM, Knaus WA, Schein RM, Sibbald WJ. Definitions for sepsis and organ failure and guidelines for the use of innovative therapies in sepsis. The ACCP/SCCM Consensus Conference Committee. American College of Chest Physicians/Society of Critical Care Medicine. Chest. 1992 Jun;101(6):1644-55. doi: 10.1378/chest.101.6.1644. PMID 1303622
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Jain S, Guleria K, Suneja A, Vaid NB, Ahuja S. Use of the Sequential Organ Failure Assessment score for evaluating outcome among obstetric patients admitted to the intensive care unit. Int J Gynaecol Obstet. 2016 Mar;132(3):332-6. doi: 10.1016/j.ijgo.2015.08.005. Epub 2015 Dec 2. PMID 26792141
- [Background] Arts DG, de Keizer NF, Vroom MB, de Jonge E. Reliability and accuracy of Sequential Organ Failure Assessment (SOFA) scoring. Crit Care Med. 2005 Sep;33(9):1988-93. doi: 10.1097/01.ccm.0000178178.02574.ab. PMID 16148470
- See also: Maternal mortality - WHO — https://www.who.int/news-room/fact-sheets/detail/maternal-mortality
- See also: Weekly Epidemiological Bulletin, number 21 of 2017 (May 21 - May 27) — https://www.ins.gov.co/buscador-eventos/BoletinEpidemiologico/2017%20Bolet%C3%ADn%20epidemiol%C3%B3gico%20semana%2021.pdf